CLINICAL TRIAL: NCT07065448
Title: The Reliability of the Elbow Isotonic Contraction Test as an Alternative to the Gait Speed Test in Assessing Sarcopenia Severity
Brief Title: Alternative to Gait Speed in Sarcopenia Assessment
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, M.D., Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPRMTRH-TYY1
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia; Elderly
Keywords: sarcopenia; reliability and validity; muscle strength; upper extremity function; physical performance parameters
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: older adults with sarcopenia
  Interventions: Other: physical performance tests
- Group 2: healthy young adults
  Interventions: Other: physical performance tests

INTERVENTIONS:
Other: physical performance tests — All participants underwent the 4-meter Gait Speed Test, the Short Physical Performance Battery (SPPB), the Timed Up and Go (TUG) test, and the Elbow Performance Test twice, with a 7-10-day interval between sessions. In the Elbow Performance Test, a 1-kilogram sandbag was fixed to the distal forearm of the dominant arm, and participants were asked to perform 30 consecutive elbow flexion-extension movements.

SUMMARY:
This study aims to assess the reliability of the Elbow Performance Test as an upper extremity-based alternative for evaluating sarcopenia severity. Unlike traditional lower extremity-focused assessments, this test may offer a practical solution for individuals with mobility limitations or comorbidities affecting the lower limbs. Participants will include older adults with sarcopenia and healthy young adults. Functional tests, including the 4-meter Gait Speed Test, SPPB, TUG, and the Elbow Performance Test, will be administered twice within a 7-10-day interval. Reliability will be analyzed using intraclass correlation coefficients (ICC).

DETAILED DESCRIPTION:
Background:Sarcopenia is a generalized and progressive skeletal muscle disorder characterized by a decline in muscle strength, mass, and function. The severity of sarcopenia is commonly assessed using functional performance tests, which are also used for monitoring disease progression and treatment response. However, lower extremity-based tests may have limited applicability in the presence of various comorbidities.

Objective: This study proposes an upper extremity-based alternative, the Elbow Performance Test, and aims to evaluate its reliability in comparison to the commonly used 4-meter Gait Speed Test.

Method:This planned cross-sectional study will include two groups: older adults with sarcopenia and healthy young adults. All participants will undergo the 4-meter Gait Speed Test, the Short Physical Performance Battery (SPPB), the Timed Up and Go (TUG) test, and the Elbow Performance Test on two separate occasions, with a 7-10-day interval between sessions. In the Elbow Performance Test, a 1-kilogram sandbag will be attached to the distal forearm of the dominant arm, and participants will be instructed to perform 30 consecutive elbow flexion-extension movements. The total time required to complete the repetitions will be recorded. The reliability of the test will be evaluated using intraclass correlation coefficients (ICC).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who consent to participate in the study

  *Sarcopenia Group
* Male participants aged 60 years or older
* Diagnosed with sarcopenia according to EWGSOP2 criteria

  *Healthy Young Control Group
* Male participants aged 40 years or younger
* SARC-F screening test score < 4

Exclusion Criteria:

* Inability to cooperate
* Poor general condition due to acute medical problems
* Chronic decompensated cardiac, renal, or hepatic failure
* Presence of rheumatologic, psychiatric, or neurological disorders
* Use of performance-enhancing or fatigue-reducing medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sarcopenia Group and Healthy Young Control Group
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
the Elbow Performance Test | Two assessment sessions conducted seven to ten days apart to evaluate test-retest reliability using intraclass correlation coefficients (ICC).
  The total time required to complete thirty consecutive elbow flexion-extension movements, performed with a one-kilogram sandbag attached to the distal forearm of the dominant arm.

SECONDARY OUTCOMES:
the 4-meter Gait Speed Test | Two assessment sessions conducted seven to ten days apart to evaluate test-retest reliability using intraclass correlation coefficients (ICC).
  The 4-Meter Gait Speed Test was used to evaluate functional mobility. Participants walked a total of 6 meters at their usual pace, with timing recorded only for the central 4-meter section. A stopwatch was used to measure the time, and gait speed was calculated in meters per second.
the Short Physical Performance Battery (SPPB) | Two assessment sessions conducted seven to ten days apart to evaluate test-retest reliability using intraclass correlation coefficients (ICC).
  Physical performance will be assessed using the Short Physical Performance Battery (SPPB), which includes balance tests (standing positions), the 4-meter gait speed test, and the five-times sit-to-stand test. Each component is scored from 0 to 4, yielding a total score ranging from 0 to 12, with higher scores indicating better physical function.
Timed Up and Go (TUG) | Two assessment sessions conducted seven to ten days apart to evaluate test-retest reliability using intraclass correlation coefficients (ICC).
  Functional mobility and balance will be assessed using the Timed Up and Go (TUG) test, which measures the time required to stand up from a chair, walk three meters, turn around, and sit back down.

CONTACTS AND LOCATIONS:
Overall Officials: İlhan Karacan, Prof., Study Director — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahat G, Tufan A, Tufan F, Kilic C, Akpinar TS, Kose M, Erten N, Karan MA, Cruz-Jentoft AJ. Cut-off points to identify sarcopenia according to European Working Group on Sarcopenia in Older People (EWGSOP) definition. Clin Nutr. 2016 Dec;35(6):1557-1563. doi: 10.1016/j.clnu.2016.02.002. Epub 2016 Feb 11. PMID 26922142
- [Background] Power GA, Dalton BH, Rice CL. Human neuromuscular structure and function in old age: A brief review. J Sport Health Sci. 2013 Dec;2(4):215-226. doi: 10.1016/j.jshs.2013.07.001. PMID 27011872
- [Background] Karacan I, Turker KS. Exploring neuronal mechanisms of osteosarcopenia in older adults. J Physiol. 2026 Jan;604(2):672-688. doi: 10.1113/JP285666. Epub 2024 Aug 9. PMID 39119811
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372